CLINICAL TRIAL: NCT00735189
Title: Does Anticoagulant Control Change Following Referral Back to the Primary Care Physician? A Prospective Randomized Trial
Brief Title: Does Anticoagulant Control Change Following Referral Back to the Primary Care Physician?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Dr. Tammy J. Bungard, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: epicore ams1
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Warfarin
Keywords: warfarin; anticoagulation; anticoagulation clinics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patient continues to receive anticoagulation care from the Anticoagulation Management Service
  Interventions: Other: anticoagulation clinic care
- 2 (Active Comparator): Patient receives anticoagulation care from their usual primary care physician
  Interventions: Other: usual care

INTERVENTIONS:
Other: anticoagulation clinic care — Patient receives care from the outpatient anticoagulation management service
  Arms: 1
Other: usual care — patient receives usual anticoagulation care from their regular primary care physician
  Arms: 2

SUMMARY:
Warfarin is a medication typically referred to as a blood thinner and is used to prevent the formation of blood clots, and hence prevent life-threatening events such as strokes and clots on the lungs (known as pulmonary emboli). This therapy is only safe and effective if the degree of blood thinning is kept within a narrow window - if the blood is "too thick" clots may form but if the blood is "too thin" the risk of bleeding increases. Complicating the control of warfarin is that different people require different amounts of it to have an appropriate degree of blood thinning, and once this amount is determined for a patient, it may be changed by factors that are encountered on a daily basis (i.e., diet, acute and chronic diseases, alcohol, medications, etc.). As such, regular monitoring is necessary to confer the benefits of this medication. Our Anticoagulation Management Service (AMS) has demonstrated really good control of blood thinning therapy by working with patients to inform them of the rationale for this medicine, the factors having the ability to impact its control, and encouraging the patient to be involved in their care (via provision of tools to document test results, one-on-one education and access to our program at any time with questions, etc.) Currently, our AMS has to limit the volume of patients seen due to resource limitations. As such, it is imperative that we investigate alternate strategies to manage these patients. Paramount, however, is that any long-term strategy must not confer inferior control of warfarin. The purpose of this study is to determine if the impact of AMS Care is sustained following the transfer of anticoagulation management to the family doctor. Operationally, the results of this study will guide future management of patients. If control of warfarin therapy declines with family doctor management, alternate strategies, such as patient self-management, will need to be investigated in a larger scale trial.

ELIGIBILITY:
Inclusion Criteria:

* current patient of the Anticoagulation Management Service
* anticipated need for long term anticoagulation
* have a regular primary care physician

Exclusion Criteria:

* previous failure of warfarin therapy (a bleed or clot despite therapeutic anticoagulation
* have a planned procedure (surgery) mandating discontinuation of warfarin
* are taking warfarin for a mechanical valve indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Adequacy of anticoagulation control (proportion of time in the therapeutic anticoagulation range +/- 0.5 INR unit) by the Rosendaal method. | 6 months

SECONDARY OUTCOMES:
Time within expanded therapeutic range (+/- 0.7 INR unit) by the Rosendaal method | 6 months
Rates of thrombosis between groups | 6 months
Rates of major hemorrhage between groups | 6 months
Patient satisfaction via postal survey | 6 months
Rate of crossover from primary care physician group back to anticoagulation management service | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tammy J Bungard, PharmD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada